CLINICAL TRIAL: NCT06287021
Title: Bone Remodeling Around a 3D-printed Highly-porous Trabecular Titanium Acetabular Cup in Primary Total Hip Arthroplasty
Brief Title: Bone Remodeling Around a Trabecular Titanium Cup in Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Permedica spa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRASERBMD2022
Record Dates: First submitted 2024-02-09; First posted 2024-02-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Total Hip Arthroplasty
Keywords: Bone Mineral Density; DEXA; Additive Manufacturing; 3D-Printing; Selective Laser Melting; Highly-Porous Titanium

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, unblinded, multicenter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jump System Traser® cup (Experimental): 25 patients receiving unilateral primary total hip arthroplasty with the Jump System Traser® acetabular cup, a 3D-printed highly-porous titanium cup
  Interventions: Device: Jump System Traser® cup
- Jump System HAX-Pore® cup (Active Comparator): 25 patients receiving unilateral primary total hip arthroplasty with the Jump System HAX-Pore® acetabular cup, a standard hydroxyapatite/titanium plasma-sprayed cup
  Interventions: Device: Jump System HAX-Pore® cup

INTERVENTIONS:
Device: Jump System Traser® cup — Press-fit, cementless, 3D-printed, highly-porous trabecular titanium acetabular cup
  Arms: Jump System Traser® cup
Device: Jump System HAX-Pore® cup — Press-fit, cementless, hydroxyapatite/titanium plasma-sprayed acetabular cup
  Arms: Jump System HAX-Pore® cup

SUMMARY:
The goal of this randomized controlled trial is to measure the periprosthetic bone mineral density changes around a 3D-printed highly-porous titanium acetabular cup used in primary total hip arthroplasty compared to a standard hydroxyapatite/titanium plasma-sprayed acetabular cup up to 2-year follow-up.

DETAILED DESCRIPTION:
In joint arthroplasty, the need to use devices with highly-porous structures even more close to cancellous bone, arises from the need of optimal implant primary stability and osseointegration to guarantee long term longevity of the prosthetic implant.

After decades of clinical use of highly-porous tantalum (Trabecular Metal) acetabular components in total hip arthroplasty with excellent results, new highly-porous titanium structures have been developed and introduced in the market thanks to the additive manufacturing technology.

This study aims to investigate how bone remodeling occurs after primary total hip arthroplasty around a highly-porous trabecular-irregular acetabular cup, 3D-printed with selective laser melting, in comparison with a standard hydroxyapatite/titanium plasma-sprayed cup with the same design. The null hypothesis, which the study aims to reject, is that there is no difference in bone mineral density changes between highly-porous and traditional plasma-sprayed cups.

Overall 50 patients will be enrolled to be 1:1 randomized for receiving the investigational cup or the control cup in two centers.

Periprosthetic bone mineral density will be measured by DEXA (Dual-Energy X-ray Absorptiometry) around the acetabular cup according to four ROI (Region Of Interest). DEXA scans will be taken at different time-points up to 2-year follow-up. DEXA scan taken before patient discharge will be used as baseline.

Patients will be assessed also for clinical and radiological results, with focus on osseointegration signs of the acetabular cup.

ELIGIBILITY:
Inclusion Criteria:

* Patient candidated to undergo unilateral cementless primary total hip arthroplasty with Jump System Traser® cup or Jump System HAX-Pore® cup by Permedica Orthopaedics (study sponsor).
* Patient with primary or secondary hip osteoarthritis;
* Patient who has given informed consent;

Exclusion Criteria:

* Male patients younger than 40 years or older than 85 years;
* Female patients younger than 50 years or older than 85 years;
* Childbearing;
* Patients not indicated for receiving the investigational devices;
* Patients not indicated for receiving cementless metaphyseal short femoral stems by Permedica Orthopaedics as the "Exacta RS" or "Exacta S" brand;
* Patients with rheumatoid arthritis, avascular osteonecrosis, severe hip dysplasia (grade III-IV according to Crowe classification), Perthes disease, Paget disease, femoral neck fracture, pelvic fracture or sequelae of previous surgical procedures or trauma to the ipsilateral hip;
* Patients with bone disorders;
* Patients with diabetes;
* Patients under PTH (parathyroid hormone), corticosteroid, or osteoporosis pharmacological therapy;
* Patients with disabling disease in the contralateral limb;
* Patients with BMI > 30 or < 18;
* Patients not willing to follow the study protocol;
* Patients incapable to understand the study protocol;
* Patients addicted to alcohol or drugs;
* Patients already enrolled in other clinical investigations;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
BMD - ROI 1 | Preoperative, 1 week postoperatively, 3-month, 6-month,12-month, and 24-month follow-up
  Periprosthetic BMD (bone mineral density) measured by DEXA in ROI (region of interest) 1 (above the acetabular cup)

SECONDARY OUTCOMES:
BMD - ROI 2,3,4 | Preoperative, 1 week postoperatively, 3-month, 6-month,12-month, and 24-month follow-up
  Periprosthetic BMD (bone mineral density) measured by DEXA in ROI (region of interest) 2, 3 and 4 (behind and below the acetabular cup)
Harris hip score | Preoperative,12-month, and 24-month follow-up
  Clinical score for hips undergoing total hip arthroplasty. The Harris hip score ranges from 0 to 100, where 100 indicates the best outcome possible for the patient.
Moore's osseointegration signs | 12-month and 24-month follow-up
  Five radiographic signs around the acetabular cup revealing the stability and osseointegration status of cementless component: (1) absence of radiolucent lines; (2) presence of a superolateral buttress; (3) medial stress-shielding; (4) radial trabeculae; and (5) an inferomedial buttress.
  The presence of 3 to 5 signs visible on anterior-posterior radiograph of the hip indicates 97% probability of a well osseointegrated cup. The presence of 1 or no signs indicates 83% probability of unstable, not osseointegrated cup.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Banci, MSc, Study Director — Permedica Orthopaedics, Merate, Italy; Giuseppe Peretti, MD, Principal Investigator — IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy; Paolo Sirtori, MD, Principal Investigator — Istituto Clinico San Siro, Milan, Italy
Locations (2):
- Italy (2):
  - IRCCS Istituto Clinico San Siro, Milan
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hemmila M, Karvonen M, Laaksonen I, Matilainen M, Eskelinen A, Haapakoski J, Puhto AP, Kettunen J, Manninen M, Makela KT. Survival of 11,390 Continuum cups in primary total hip arthroplasty based on data from the Finnish Arthroplasty Register. Acta Orthop. 2019 Aug;90(4):312-317. doi: 10.1080/17453674.2019.1603596. Epub 2019 Apr 17. PMID 30994043
- [Background] Paxton EW, Mohaddes M, Laaksonen I, Lorimer M, Graves SE, Malchau H, Namba RS, Karrholm J, Rolfson O, Cafri G. Meta-analysis of individual registry results enhances international registry collaboration. Acta Orthop. 2018 Aug;89(4):369-373. doi: 10.1080/17453674.2018.1454383. Epub 2018 Mar 28. PMID 29589467
- [Background] Laaksonen I, Lorimer M, Gromov K, Eskelinen A, Rolfson O, Graves SE, Malchau H, Mohaddes M. Trabecular metal acetabular components in primary total hip arthroplasty. Acta Orthop. 2018 Jun;89(3):259-264. doi: 10.1080/17453674.2018.1431445. Epub 2018 Feb 5. PMID 29400118
- [Background] Macheras GA, Lepetsos P, Leonidou AO, Anastasopoulos PP, Galanakos SP, Poultsides LA. Survivorship of a Porous Tantalum Monoblock Acetabular Component in Primary Hip Arthroplasty With a Mean Follow-Up of 18 Years. J Arthroplasty. 2017 Dec;32(12):3680-3684. doi: 10.1016/j.arth.2017.06.049. Epub 2017 Jul 6. PMID 28734611
- [Background] Bondarenko S, Dedukh N, Filipenko V, Akonjom M, Badnaoui AA, Schwarzkopf R. Comparative analysis of osseointegration in various types of acetabular implant materials. Hip Int. 2018 Nov;28(6):622-628. doi: 10.1177/1120700018759314. Epub 2018 May 9. PMID 29742946
- [Background] Massari L, Bistolfi A, Grillo PP, Borre A, Gigliofiorito G, Pari C, Francescotto A, Tosco P, Deledda D, Ravera L, Causero A. Periacetabular bone densitometry after total hip arthroplasty with highly porous titanium cups: a 2-year follow-up prospective study. Hip Int. 2017 Nov 21;27(6):551-557. doi: 10.5301/hipint.5000509. Epub 2017 Jul 1. PMID 28708200
- [Background] Salemyr M, Muren O, Eisler T, Boden H, Chammout G, Stark A, Skoldenberg O. Porous titanium construct cup compared to porous coated titanium cup in total hip arthroplasty. A randomised controlled trial. Int Orthop. 2015 May;39(5):823-32. doi: 10.1007/s00264-014-2571-z. Epub 2014 Oct 22. PMID 25338110
- [Background] Lazarinis S, Milbrink J, Mattsson P, Mallmin H, Hailer NP. Bone loss around a stable, partly threaded hydroxyapatite-coated cup: a prospective cohort study using RSA and DXA. Hip Int. 2014 Mar-Apr;24(2):155-66. doi: 10.5301/hipint.5000104. Epub 2014 Feb 3. PMID 24500826
- [Background] Periasamy K, Watson WS, Mohammed A, Murray H, Walker B, Patil S, Meek RM. A randomised study of peri-prosthetic bone density after cemented versus trabecular fixation of a polyethylene acetabular component. J Bone Joint Surg Br. 2011 Aug;93(8):1033-44. doi: 10.1302/0301-620X.93B8.26233. PMID 21768625
- [Background] Baad-Hansen T, Kold S, Nielsen PT, Laursen MB, Christensen PH, Soballe K. Comparison of trabecular metal cups and titanium fiber-mesh cups in primary hip arthroplasty: a randomized RSA and bone mineral densitometry study of 50 hips. Acta Orthop. 2011 Apr;82(2):155-60. doi: 10.3109/17453674.2011.572251. Epub 2011 Mar 25. PMID 21434845
- [Background] Meneghini RM, Ford KS, McCollough CH, Hanssen AD, Lewallen DG. Bone remodeling around porous metal cementless acetabular components. J Arthroplasty. 2010 Aug;25(5):741-7. doi: 10.1016/j.arth.2009.04.025. Epub 2009 May 26. PMID 19473807
- [Background] Laursen MB, Nielsen PT, Soballe K. Bone remodelling around HA-coated acetabular cups : a DEXA study with a 3-year follow-up in a randomised trial. Int Orthop. 2007 Apr;31(2):199-204. doi: 10.1007/s00264-006-0148-1. Epub 2006 Jun 8. PMID 16761153
- [Background] Digas G, Karrholm J, Thanner J. Different loss of BMD using uncemented press-fit and whole polyethylene cups fixed with cement: repeated DXA studies in 96 hips randomized to 3 types of fixation. Acta Orthop. 2006 Apr;77(2):218-26. doi: 10.1080/17453670610045948. PMID 16752282
- [Background] Ragone V, Canciani E, Arosio M, Olimpo M, Piras LA, von Degerfeld MM, Augusti D, D'Ambrosi R, Dellavia C. In vivo osseointegration of a randomized trabecular titanium structure obtained by an additive manufacturing technique. J Mater Sci Mater Med. 2020 Jan 21;31(2):17. doi: 10.1007/s10856-019-6357-0. PMID 31965345